CLINICAL TRIAL: NCT01610024
Title: Northern Board Beet Breathlessness Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Health and Social Care Trust (Other Government)
Responsible Party: Principal Investigator, Dr. Wendy Anderson, Consultant Respiratory Physician, Northern Health and Social Care Trust
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: RDF001
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Exercise Tolerance (Measured in Minutes)

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Beetroot (Active Comparator)
  Interventions: Dietary Supplement: Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — Give subjects 500ml beetroot juice in the 24 hour period prior to class begins. They will receive this during 3 of the 6 weeks

SUMMARY:
Hypothesis: Beetroot juice increases the exercise tolerance of patients with chronic lung disease.

Using the already established pulmonary rehabilitation model, we aim to split the group of 8 into 2 groups, each group taking 500ml of beetroot juice 24 hours before there class on alternate (differing) weeks to see if it improves their overall exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Already planned to attend the pulmonary rehabilitation class

Exclusion Criteria:

* Angina Prescribed regular nitrates, a resting heart rate >100bpm, a resting blood pressure <110 systolic, postural hypotension, prescribed PDE5 inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Exercise Tolerance | 6 weeks
  Measuring incremental change in exercise tolerance between weeks of beetroot consumption and weeks of no beetroot consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Antrim Area Hospital, Antrim, County Antrim, United Kingdom